CLINICAL TRIAL: NCT01332669
Title: Multicenter Registry of Chemoembolization Using Drug-eluting Bead in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Drug-eluting Bead in Hepatocellular Carcinoma
Acronym: REDEBUT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin Wook Chung, professor of radiology, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Biocompatible-Korea
Record Dates: First submitted 2011-02-06; First posted 2011-04-11 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; chemoembolization; drug eluting beads; HCC; Liver cancer; Korea
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chemoembolization (Active Comparator): HCC patients received chemoembolization
  Interventions: Procedure: DebDox TACE
- Historical use of c-TACE using Lipiodiol and doxorubicin (Other): The control arm will be of the patients that have been treated historically in the centers with conventional TACE (that is Lipiodiol plus doxorubicin).
  Interventions: Procedure: DebDox TACE

INTERVENTIONS:
Procedure: DebDox TACE — HCC patients will receive chemoembolization (TACE) using DC beads containing Doxorubicin. The objective is to give 2 vials of DC Bead (2ml per vial) loaded with 70-75mg of Doxorubicin per vial (Each vial contain 2ml of DC Bead, thus doxorubicin concentration will be of 35-37.5mg per ml of DC Beads)
  Other Names: chemoembolization using drug eluting beads; DC bead chemoembolization; DebDox; TACE

SUMMARY:
In unresectable hepatocellular carcinoma, TACE using Lipiodol/anti cancer agent emulsion is the standard treatment and reported as a significantly better treatment through randomized comparison study like Llovet, etc. than conservative treatment. Recently, doctors do transarterial chemoembolization with drug-eluting bead, and it is proved less side effect and better efficacy than conventional TACE using Lipiodol in Precision V study by Dr. Lammer, etc. But, it could not defined improved survival rate as expected. This study's purpose is evaluating treatment efficacy, survival rate and safety of TACE using drug eluting bead by comparing to conventional TACE using doxorubicin/Lipiodol emulsion for unresectable hepatocellular carcinoma.

DETAILED DESCRIPTION:
Comparison Between Drug-Eluting Bead vs conventional TACE.

Drug-eluting bead group : TACE using DC bead loading Doxorubicin. Conventional TACE group : TACE using Doxorubicin/Lipiodol emulsion and gelatin sponge/PVA particle.

cTACE group was chosen by concurrent matched patients (age, sex, tumor stage, and Child-Pugh class are matched)

5.7 Technically considerable aspects of DC bead TACE group

1. Planned dose of doxorubicin. Each vial of DC Bead (2 ml of beads) should be loaded with 70-75 mg doxorubicin (loading dose, 35-37.5 mg doxorubicin / ml of beads).

   * Early-stage HCC. As a general rule, each single treatment should include a planned dose of up to 75 mg doxorubicin loaded into one vial of DC Bead.
   * Medium-sized (less than 8cm) / multinodular HCC. As a general rule, each single treatment should include a planned dose of up to 150 mg doxorubicin loaded into two vials of DC Bead.
   * In large tumors (more than 8cm), even if unilobar, the separate treatment including two sessions 2-4 weeks apart is recommended.
   * In bilobar tumors, both hepatic lobes should be treated in separate treatment sessions 2-4 weeks apart, in the absence of complications requiring a longer time interval between the two sessions. Obtaining confirmation that the liver enzymes did return to baseline before performing the second treatment session is recommended.
2. Choice of DC Bead size. Use of 100-300μm beads is recommended for a standard procedure. However, individual patient and tumor characteristics, particularly the identification of arterio-venous shunting, should be taken into account when the safety of the treatment and the choice of DC Bead size are determined.

   * In the case of significant arterio-portal or hepatic venous shunting, embolization of the shunt with gelfoam pledgets is recommended before proceeding with DEBDOX. Confirmation that the shunt is no longer present must be obtained before DEBDOX can safely be performed. But, this study excludes the patients with arterio-portal or hepatic venous shunts.
   * In large tumors, hepatic arterial flow does not reach 'near stasis' after injection of 2 vial of 100-300 μm DC beads. The recommendation is following: 2 vials of the 100-300 μm DC beads is best and then repeat 2 weeks later if the patient is doing well clinically.
3. DC Bead dilution. Mix loaded DC Bead with a non-ionic contrast medium. At least 5-10 ml of non-ionic contrast should be used per 1 ml of DC Bead (i.e., 10-20 ml are required to dilute one vial of DC Bead) prior to injection.
4. Catheter positioning. A superselective (i.e., segmental or subsegmental) approach should be used whenever possible by using a microcatheter. Use of 3D / MPR obtained from C-arm rotational angiography with a flat-panel detector system (cone-beam CT) is recommended, if available, to improve the accuracy in identifying tumor-feeding arteries. Such imaging allows for accurate targeting of the tumor. In addition, repeat cone beam CT should be performed after successful delivery of the DC Bead to confirm adequate targeting and saturation of the tumor(s).

   * Segmental / subsegmental approach. Place the microcatheter into the segmental / subsegmental vessel feeding the tumor as distally as possible - but avoiding wedging the catheter to avoid reflux along the catheter shaft. Flow within the artery must be preserved.
   * Lobar approach. Place the catheter as selectively as possible in the right or left hepatic artery. Pay attention to identifying the origin of the cystic artery as well as other arteries supplying flow to extra-hepatic organs such as the right gastric artery, para-esophageal or omental vessels among others. If identified, these vessels must be either embolized using coils or avoided by placing the catheter tip well beyond the origin of these vessels. In addition, forward flow into the desired vessel must be maintained as inadvertent administration of even a few DC Beads into these extra-hepatic vessels could have dire consequences.
5. Injection. The injection must be very slow. An injection rate of 1 ml of the contrast agent - DC Bead suspension per minute is recommended. Thus, it takes 10-20 minutes to infusion 1 vial of DC bead. Care should be taken to avoid sedimentation of the beads in the syringe by rotating the syringes or using a 3-way stopcock to gently suspend the beads in the solution.
6. Embolisation endpoint. Injection should be continued until "near stasis" is observed in the artery directly feeding the tumor (i.e., the contrast the contrast column should clear within 2-5 heart beats). At that point, injection should be stopped - regardless of the amount of beads that have been actually administered - to avoid reflux of embolic material. Once the embolisation endpoint has been achieved, no additional embolic material should be injected. If the "near stasis" endpoint is not obtained after injection of the scheduled volume of beads, no additional embolization should be performed. This patient is likely to benefit from a second course after imaging follow-up.
7. extrahepatic collateral vessels. In principle, DC bead is used for collateral arterial circulation (inferior phrenic artery, internal mammary artery, intercostal artery), but doctors can do bland embolization (PVC particle, gelatin sponge) based on their judgement.
8. Repeated treatment. In principle, treatment with the same method is repeated for every 2 - 3 months as tumor progression is observed. But, even if tumor progression is not observed, the treatment can be repeated for tumor repression. If there is no tumor left, contrast enhancement CT or MRI can be performed for every 2- 3 months as follow up.

5.8. Dose in study Dose of DC bead, anti cancer agent for TACE dose is decided by tumor size. So, this study just set up the maximum dose.

Drug-eluting bead group DC bead : 2 bottles DC bead absorbs 70-75mg per bottle. Doxorubicin loading to DC bead needs to be done 1.5 hours before using. The size of DC bead is 100-300 micrometer, and it can be used up to 2 bottles.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed diagnosis of HCC as stated below

   * Cirrhotic subjects: Clinical diagnosis by AASLD criteria
   * Non-cirrhotic subjects: histological confirmation is mandatory
2. Patient with HCC not suitable for radical therapies such as resection, liver transplantation or percutaneous therapies or patient is indicated for these therapies but there is a contraindication for them or patient himself rejects above treatments and wants to do TACE (Indication for hepatectomy, liver transplantation, local ablation is decided by doctors of each center)
3. Multinodular or single nodular tumor over 5cm, (In the case of single nodule less than 5cm, if curative treatment is contraindicated or the patient rejects curative treatment)
4. Hypervascular lesion showing contrast enhancement in the early stage at the contrast media bolus injection CT or MRI.
5. At least one uni-dimensional lesion measurable according to the Modified RECIST criteria by CT-scan or MRI
6. No invasion in the blood vessel (hepatic portal, hepatic vein) or bile duct by the CT or MR
7. Eastern Cooperative Oncology Group performance status is 0 - 1
8. Child-Pugh classification is A or B7
9. Proper blood, liver, renal, heart function: testing result within 2 weeks from registry of this study is followed:

   * white blood cell number : > 3,000/mm2
   * platelet number : > 5 x 104/mm3
   * blood bilirubin : < 3.0 mg/dL
   * ASL, ALT is within 5 times of normal range of each organ
   * serum creatinine : < 1.5 mg/dL
   * hemoglobin : > 8.0 g/dL
10. Over 20 years old
11. Expected survival more than 6 months
12. Patients who are willing to do regular visit, laboratory test, and radiological exam
13. Prior written patient consent

Exclusion Criteria:

1. ECOG performance status 2 or more, Child-Pugh class B8 or more
2. Diffuse HCC or presence of vascular or biliary invasion or extrahepatic spread.
3. Vascular or biliary invasion
4. Extrahepatic metastasis (Any lymph nodes measuring ≥ 10mm along the short axis)
5. Tumor burden involving more than 50% of the liver
6. Patients previously treated with any anti-cancer therapy for HCC except hepatic resection or early recurrence within 1 year after resection
7. Liver cancer rupture
8. History of biliary tract repair or endoscopic biliary tract treatment
9. Clinically important refractory ascites or pleural fluid
10. Any contraindications for hepatic embolization procedures

    * Known hepatofugal blood flow
    * Arterio-venous shunt
    * Impaired clotting test (platelet count < 5 x 104/mm3, PT-INR > 2.0)
11. Any contraindication for doxorubicin administration
12. Contrast media allergy contraindicating angiography
13. Acute or active following diseases

    * Heart failure can't control, angina pectoris and/or arrhythmia diseases
    * Myocardial infarction within the last 6months,
    * Renal failure
    * Active infection (virus infection can be accepted)
    * Active hemorrhage of digestive system
    * Other malignant tumor history
    * Hepatic coma or acute mental disease
14. Pregnant, nursing or childbearing age women and men who are actively sexually available and don't want to or can't do contraception
15. Safety concerns based on researcher's judge

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
tumor response | 6 months

SECONDARY OUTCOMES:
survival rate | 2 years
Incidence rate and grade of side effect | 6months
Time to progression | 2 years
Time to untreatable progression | 2 years
Number of treatment required to achieve objective response | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jin Wook Chung, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Dhanasekaran R, Kooby DA, Staley CA, Kauh JS, Khanna V, Kim HS. Comparison of conventional transarterial chemoembolization (TACE) and chemoembolization with doxorubicin drug eluting beads (DEB) for unresectable hepatocelluar carcinoma (HCC). J Surg Oncol. 2010 May 1;101(6):476-80. doi: 10.1002/jso.21522. PMID 20213741
- [Background] Malagari K, Pomoni M, Kelekis A, Pomoni A, Dourakis S, Spyridopoulos T, Moschouris H, Emmanouil E, Rizos S, Kelekis D. Prospective randomized comparison of chemoembolization with doxorubicin-eluting beads and bland embolization with BeadBlock for hepatocellular carcinoma. Cardiovasc Intervent Radiol. 2010 Jun;33(3):541-51. doi: 10.1007/s00270-009-9750-0. Epub 2009 Nov 24. PMID 19937027
- [Background] Malagari K, Pomoni M, Spyridopoulos TN, Moschouris H, Kelekis A, Dourakis S, Alexopoulou E, Koskinas J, Angelopoulos M, Kornezos J, Pomoni A, Tandeles S, Marinis A, Rizos S, Kelekis D. Safety profile of sequential transcatheter chemoembolization with DC Bead: results of 237 hepatocellular carcinoma (HCC) patients. Cardiovasc Intervent Radiol. 2011 Aug;34(4):774-85. doi: 10.1007/s00270-010-0044-3. Epub 2010 Dec 24. PMID 21184228
- [Background] Nicolini A, Martinetti L, Crespi S, Maggioni M, Sangiovanni A. Transarterial chemoembolization with epirubicin-eluting beads versus transarterial embolization before liver transplantation for hepatocellular carcinoma. J Vasc Interv Radiol. 2010 Mar;21(3):327-32. doi: 10.1016/j.jvir.2009.10.038. Epub 2010 Jan 22. PMID 20097098
- [Background] Poon RT, Tso WK, Pang RW, Ng KK, Woo R, Tai KS, Fan ST. A phase I/II trial of chemoembolization for hepatocellular carcinoma using a novel intra-arterial drug-eluting bead. Clin Gastroenterol Hepatol. 2007 Sep;5(9):1100-8. doi: 10.1016/j.cgh.2007.04.021. Epub 2007 Jul 12. PMID 17627902
- [Background] Lammer J, Malagari K, Vogl T, Pilleul F, Denys A, Watkinson A, Pitton M, Sergent G, Pfammatter T, Terraz S, Benhamou Y, Avajon Y, Gruenberger T, Pomoni M, Langenberger H, Schuchmann M, Dumortier J, Mueller C, Chevallier P, Lencioni R; PRECISION V Investigators. Prospective randomized study of doxorubicin-eluting-bead embolization in the treatment of hepatocellular carcinoma: results of the PRECISION V study. Cardiovasc Intervent Radiol. 2010 Feb;33(1):41-52. doi: 10.1007/s00270-009-9711-7. Epub 2009 Nov 12. PMID 19908093
- [Background] Takayasu K, Arii S, Ikai I, Omata M, Okita K, Ichida T, Matsuyama Y, Nakanuma Y, Kojiro M, Makuuchi M, Yamaoka Y; Liver Cancer Study Group of Japan. Prospective cohort study of transarterial chemoembolization for unresectable hepatocellular carcinoma in 8510 patients. Gastroenterology. 2006 Aug;131(2):461-9. doi: 10.1053/j.gastro.2006.05.021. PMID 16890600
- [Background] Llovet JM, Di Bisceglie AM, Bruix J, Kramer BS, Lencioni R, Zhu AX, Sherman M, Schwartz M, Lotze M, Talwalkar J, Gores GJ; Panel of Experts in HCC-Design Clinical Trials. Design and endpoints of clinical trials in hepatocellular carcinoma. J Natl Cancer Inst. 2008 May 21;100(10):698-711. doi: 10.1093/jnci/djn134. Epub 2008 May 13. PMID 18477802
- [Background] Bruix J, Sherman M; Practice Guidelines Committee, American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma. Hepatology. 2005 Nov;42(5):1208-36. doi: 10.1002/hep.20933. No abstract available. PMID 16250051
- [Background] Varela M, Real MI, Burrel M, Forner A, Sala M, Brunet M, Ayuso C, Castells L, Montana X, Llovet JM, Bruix J. Chemoembolization of hepatocellular carcinoma with drug eluting beads: efficacy and doxorubicin pharmacokinetics. J Hepatol. 2007 Mar;46(3):474-81. doi: 10.1016/j.jhep.2006.10.020. Epub 2006 Nov 29. PMID 17239480
- [Background] Llovet JM, Real MI, Montana X, Planas R, Coll S, Aponte J, Ayuso C, Sala M, Muchart J, Sola R, Rodes J, Bruix J; Barcelona Liver Cancer Group. Arterial embolisation or chemoembolisation versus symptomatic treatment in patients with unresectable hepatocellular carcinoma: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1734-9. doi: 10.1016/S0140-6736(02)08649-X. PMID 12049862
- See also: efficacy of DEB in chemoembolization of HCC — http://www.projectsinknowledge.com/
- See also: interventional treatment of HCC — http://www.medscape.com/